CLINICAL TRIAL: NCT02845427
Title: Closed Suction Drain or Not After Total Hip Arthroplasty: A Randomized Controlled Trial
Brief Title: Closed Suction Drain or Not After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yasser E khalifa, professor doctor of orthopedic and traumatology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUHOR1
Record Dates: First submitted 2016-07-14; First posted 2016-07-27 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2017-02

CONDITIONS: Total Hip Arthroplasty
Keywords: Closed Suction Drain; Wound Hematoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A(drain group) (Active Comparator): patients of primary THA will have closed suction drain introduced intraoperative at surgical site
  Interventions: Device: closed suction drain
- B(No drain group) (Placebo Comparator): patients of primary THA will have the surgical wound be closed with no suction drain
  Interventions: Procedure: no suction drain

INTERVENTIONS:
Device: closed suction drain — using closed suction drain system postoperative
  Arms: A(drain group)
Procedure: no suction drain — the surgical wound will be closed with no suction drain
  Arms: B(No drain group)

SUMMARY:
Comparative randomised study to clarify which better to use or no use of closed suction drain system after total hip arthroplasty regarding amount of blood loss, need for blood transfusion, risk for superficial infection, ecchymosis, wound discharge, effect on early post-operative rehabilitation. Patients will be followed up for one month postoperative clinically (Harris Hip score system), laboratory (Hb level), and radiologically (A-P view plain x-ray of the hip).

DETAILED DESCRIPTION:
Total Hip Arthroplasty (THA) wounds are prone to formation of hematomas. Hematomas may increase the incision tension, leading to wound discharge and providing a good medium for bacteria, increase post-operative pain, limitation of range of motion of hip joint and prolong post-operative rehabilitation duration, also may cause ecchymosis, and tension vesicles around the surgical wound.

So use of closed suction drain system may reduce these complications. Nevertheless some recent studies have claimed that drainage can cause other complications and does not reduce hematoma formation and risk for infection. Furthermore, some studies have shown that drainage increase blood loss after THA which may both lead to increase blood transfusion requirements and provide an entry point for skin microorganisms.

Some other studies have found that no significance between use and non use of suction drain after THA.

So the investigators will take this issue for study a comparison between benefits and hazards of use and non use of suction drain after THA.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip arthroplasty (THA)

Exclusion Criteria:

* Revision cases
* Uncontrolled bleeding tendency (prothrombin conc. Less than 70%)
* History of deep venous thrombosis
* Sever liver impairment (liver failure)
* Sever renal impairment (S. creatinine more than 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02; Primary Completion 2017-08 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
change in Hb level | preoperative and 24 hrs postoperative

SECONDARY OUTCOMES:
amount of blood loss | upto 24 hrs postoperative
amount of blood transfusion | upto 24 hrs postoperative

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided